CLINICAL TRIAL: NCT05204043
Title: Peter Hess® Sound Massage Versus Music Care® Relaxation for the Management of Anxiety and Pain in Patients Undergoing Coronary Artery Bypass Surgery in Thoracic and Cardiovascular Surgery: a Comparative Controlled and Randomised Study.
Brief Title: Peter Hess® Sound Massage for Reducing Anxiety and Pain in Cardiac Surgery
Acronym: MuSoCa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: APHP190384; 2020-A02371-38 (Other: ANSM)
Record Dates: First submitted 2021-12-20; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Pain; Pain, Postoperative; Pain, Chest; Anxiety; Anxiety Postoperative; Thoracic Surgery
Keywords: Peter Hess; Music Care; Sound massage; sound therapy; music therapy; singing bowls; vibrations; relaxation; coronary bypass; cardiac surgery; cardiology; music
MeSH Terms: conditions — Pain; Pain, Postoperative; Chest Pain; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peter Hess® sound massage (Experimental): Peter Hess® sound massage using bowls dedicated to this technique.
  Interventions: Other: Peter Hess® sound massage; Other: Questionnaires
- Music relaxation Music Care® (Experimental): The patient chooses his music preferences and receive the music relaxation.
  Interventions: Other: Music relaxation Music Care®; Other: Questionnaires

INTERVENTIONS:
Other: Peter Hess® sound massage — The Peter Hess® sound massage uses sound vibrations generated by therapeutic singing bowls. Peter Hess' methods act far from a traumatised area, far from the pain. It will be given on the patient's bed for 30 minutes.
  Arms: Peter Hess® sound massage
Other: Music relaxation Music Care® — The patient chooses his music preferences and receive the music relaxation in bed for 30 minutes.
  Arms: Music relaxation Music Care®
Other: Questionnaires — * State Trait Anxiety Inventory (STAI)
  * Pain assessment - Visual Analogic Scale (from 0 to 10).

SUMMARY:
Cardiac surgery patients often undergo anxiousness and pain. Before surgery, anxiety is often caused by the idea of sternotomy, extracorporeal circulation, fear of post-operative pain, and even death. After surgery anxiety and pain can be the consequences of operative and peri-operative procedures. The investigators believe that reducing stress and pain by a relaxation therapy would lead to better stay in hospital and a better recovery after surgery.

Music Care® relaxation technique consists into listening to an audio relaxing soundtrack chosen by the patient. This technique has already proven with several clinical studies its efficiency for reducing pain and anxiety in hospital.

The research consists of comparing this technique to Peter Hess® sound massage for reducing pain and anxiety.

The Peter Hess® sound massage is a holistic relaxation technique that uses sound vibrations generated by therapeutic singing bowls.

Patients will be randomized in one of the two groups (Music Care® or Peter Hess®).

DETAILED DESCRIPTION:
* Cardiac surgery patients often undergo anxiousness and pain. Before surgery, anxiety is often caused by the idea of sternotomy, extracorporeal circulation, fear of post-operative pain, and even death. After surgery anxiety and pain can be the consequences of operative and peri-operative procedures. The investigators believe that reducing stress and pain by a relaxation therapy would lead to better stay in hospital and a better recovery after surgery.
* Design of the study: Controlled randomized single blind clinical trial / Interventional research protocol implying human being that doesn't involve any health product
* Patients will be randomized in one of the two following groups:

  1. Peter Hess® sound massage, a relaxation technic using singing bowls' sound vibrations The Peter Hess® sound massage is a holistic relaxation technique (body and mind) that uses sound vibrations generated by therapeutic singing bowls. Its efficiency and adaptability make it a complementary method that can be pertinent for many hospital departments, both for patients and caregivers.
  2. Music Care® relaxation technique, a validated Non-Medicinal Intervention which is a pyscho-musical relaxation technique using audio relaxation music diffused in dedicated headphone. The audio relaxing soundtracks are chosen by the patient. Music Care® technique has already proven with several clinical studies its efficiency for reducing pain and anxiety in hospital.
* Main Objective: Prove a better efficiency of the Peter Hess® sound massage for reducing anxiety compared to Music Care® relaxation technique.
* Main criteria: difference between the two groups on anxiety scores' variation (measured by STAI) between preoperative visit (J-1) and postoperative visit (J+7)

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 40 and 70 years old
2. Hospitalized for a coronary bypass
3. That has given his written consent
4. Affiliated to a French social security system or entitled to a social security benefit.

Exclusion Criteria:

1. Emergency coronary bypass surgery
2. Impaired ventricular function (ejection fraction < 45%)
3. Combined surgery
4. Patient with chronic dialysis
5. Diagnosed with severe depression
6. Patient in a psychotic state
7. Patient with chronic pain
8. Patient incapable of giving his written consent
9. Patient deprived of liberty by judicial decision or benefiting from legal protection (under guardianship or curatorship)
10. Patient on AME
11. Participation in other interventional research involving humans, or being in the period of exclusion from previous research involving humans, if applicable.
12. Pregnant or breastfeeding woman
13. Patient with pacemaker
14. Patient with implanted metallic medical devices
15. Recently operated patient
16. Patient with hearing epilepsy
17. Tinnitus patient

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory (STAI-A) score, between the 2 groups of patients | At Day7 (after surgery)
  Questionnaire based on a 4-point Likert scale and composed of 20 questions on a self-report basis.
  Higher scores are correlated with higher levels of anxiety.

SECONDARY OUTCOMES:
State Trait Anxiety Inventory (STAI-A) score, in each group | At Day-1 (day before surgery) and after surgery (at Day2 and Day4)
  Questionnaire based on a 4-point Likert scale and composed of 20 questions on a self-report basis.
  Higher scores are correlated with higher levels of anxiety.
Consumption of anxiolytic drugs | Through study completion, an average of 7 days
  Drugs prescriptions will be reported
Pain assessment | At Day-1, Day2, Day3, Day4 and Day7.
  Visual Analogic Scale (score from 0 to 10). Higher scores are correlated with higher levels of pain.
  VAS filled twice at Day-1, Day2 and Day4 (before and after the intervention (Peter Hess sound massage / Music Care)) VAS filled once at Day3 and Day7
Consumption of antalgics | Through study completion, an average of 7 days
  Drugs prescriptions will be reported
Consumption of anti-inflammatory | Through study completion, an average of 7 days
  Drugs prescriptions will be reported
Demand of care in physiotherapy | Through study completion, an average of 7 days
  Number of care in physiotherapy will be reported
Blood pressure | At Day-1 (day before surgery) and after surgery (at Day2 and Day4)
  Variation of blood pressure before and after Peter Hess sound massage or Music Care relaxation technique (depending of the arm) will be assessed
Cardiac frequency | At Day-1 (day before surgery) and after surgery (at Day2 and Day4)
  Variation of cardiac frequency before and after Peter Hess sound massage or Music Care relaxation technique (depending of the arm) will be assessed
Length of hospitalisation | At Day7 (end of participation)
  Length of hospitalisation
Sides effect | Through study completion, an average of 7 days
  Side effect reporting

CONTACTS AND LOCATIONS:
Overall Officials: Pascal LEPRINCE, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris